# **Cirrhosis Medical Home**

Eric Orman, MD
Division of Gastroenterology and Hepatology
702 Rotary Circle, Suite 225
Indianapolis, IN 46202

Co-investigators:
Malaz Boustani, MD
Noll Campbell, PharmD, MS
Nicole Fowler, PhD
Archita Desai, MD

**Support Provided by:**NIDDK

Version Date: October 4, 2021 

#### **Table of Contents:**

# **Study Schema**

- 1.0 Background & Rationale
- 2.0 Objective(s)
  - 2.1 Primary Objective
  - 2.2 Secondary Objective
- 3.0 Study Measures
  - 3.1 Primary Outcome Measure
  - 3.2 Secondary Outcome Measures
  - 3.3 Other Patient Measures
  - **3.4 Other Caregiver Measures**
- 4.0 Eligibility Criteria
  - 4.1 Patients
  - 4.2 Caregivers
- 5.0 Study Design
- 6.0 Enrollment/Randomization
- 7.0 Study Procedures
- 8.0 Study Personnel
- 9.0 Data Safety Monitoring
- 10.0 Study Withdrawal/Discontinuation
- 11.0 Statistical Considerations
- 12.0 Data Management
- 13.0 Privacy/Confidentiality Issues
- 14.0 Follow-up and Record Retention
- 15.0 References
- 16.0 Appendices
  - 16.1 Schedule of Events
  - **16.2 Sample Care Plan**

# 1.0 Background & Rationale

Every year, 150,000 Americans are hospitalized for complications of liver cirrhosis.<sup>2</sup> These patients suffer from debilitating symptoms (ascites, gastrointestinal bleeding, infection, and hepatic encephalopathy).<sup>3</sup> They also have impairments in physical, cognitive, psychological, and social functions leading to poor quality of life and long-term disability.<sup>1, 4-7</sup> These impairments contribute to high utilization of health care resources; within 30 days of hospital discharge, 25% of patients are readmitted, and of these readmissions, 20-40% are preventable.<sup>8-10</sup> This inpatient health care utilization is the largest driver of the \$30 billion spent annually on chronic liver disease.<sup>11</sup> These individual and societal burdens of cirrhosis could be improved with existing health care services, behavioral care, rehabilitation services, and community resources; but the current fragmented nature of the health care system does not allow for the necessary coordination to best care for this population.<sup>12</sup>

To address the health care system's lack of care coordination, the Institute of Medicine and Centers for Medicare and Medicaid Services recommend the development of collaborative care models (CCM) in a wide range of clinical settings.<sup>13, 14</sup> CCMs are intended to provide coordinated, personalized care pragmatically using care coordinators. CCMs have successfully improved care in multiple patient populations, ranging from frail older adults to depression.<sup>15-25</sup> In contrast, for patients with cirrhosis, there is a paucity of data to support the benefit of CCM in this medically complex and vulnerable population.<sup>26</sup> At Indiana University, researchers have over 20 years of experience in developing, testing, and implementing CCMs successfully for patients living with dementia or depression.<sup>15, 16</sup> Building on these successes, we have customized the CCM to best meet the unique and complex biopsychosocial needs of patients with cirrhosis: the Cirrhosis Medical Home.

In the Cirrhosis Medical Home, a care coordinator, supported by an interdisciplinary clinical team, will deliver a personalized intervention guided by a set of innovative tools: (i) patient-centered care protocols, (ii) a mobile office, (iii) care coordination support software, and (iv) dynamic feedback measures. The overall goal is to improve quality of life and to reduce acute health care utilization for patients with cirrhosis. In this pilot, randomized trial of 40 patients, we aim to refine our study processes in preparation for a large scale randomized controlled trial evaluating the efficacy of the Cirrhosis Medical Home in improving the quality of life of patients discharged from the hospital with cirrhosis. Additionally, up to 40 caregivers will be enrolled in the trial.

# 2.0 Objective(s)

- 2.1 The primary objective of this trial is to test the screening and enrollment processes for a randomized controlled trial of the Cirrhosis Medical Home compared to usual care for patients with decompensated cirrhosis and poor quality of life when discharged from the hospital
- **2.2** Secondary objectives are:

2.2.1 to assess the data collection process, outcome assessment, and the acceptability of the Cirrhosis Medical Home trial

2.2.2 to estimate the effect size of the Cirrhosis Medical Home intervention on quality of life at six months post hospital discharge

# 3.0 Study Measures

All primary and secondary outcomes measures will be obtained from study participants at baseline and at 3 and 6 months, per the schedule of events. Additionally, MELD and Child-Pugh scores will also be obtained at the 3 and 6 month assessments.

# 3.1 Primary Outcome (Feasibility) Measures

- **3.1.1. Enrollment rate:** The enrollment rate is the number of patients/caregivers enrolled per month. We will further determine the number of patients/caregivers screened and approached for enrollment. Based on these numbers, we will calculate the proportion of screened patients/caregivers eligible for enrollment, the proportion of eligible patients/caregivers approached, and the proportion of approached patients/caregivers enrolled. Of those not eligible, we will record reasons for ineligibility. Of those eligible, but not approached, we will record reasons. For those approached, but not enrolled, we will record reasons. **3.1.2 Drop-out rate:** The drop-out rate is the proportion of enrolled
- **3.1.2 Drop-out rate:** The drop-out rate is the proportion of enrolled participants (patients and caregivers) who drop out of the study before completion.
- **3.1.3 Data completion:** We will record the completeness of the data collection for enrolled subjects. For those with incomplete data, we will record reasons that data could not be collected.

### 3.2 Secondary Outcome Measures

- **3.2.1. Quality of Life:** This outcome will be obtained from the patient only. Patient health–related QOL will be assessed using the Medical Outcome Study Short Form (SF-36).<sup>40, 48, 49</sup> This scale has eight components (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) that are aggregated into a Physical Component Summary (PCS) and a Mental Component Summary (MCS). Changes that differ by 2 or more points on a scale of 0 to 100 are clinically meaningful.<sup>49</sup>
- **3.2.2 Physical Performance:** Physical performance measures will be obtained from the patient only. Physical recovery will be assessed via the Short Physical Performance Battery (SPPB), a validated objective assessment. The SPPB yields a performance score of 0-12 (0-4 poor, 5-7 intermediate, 8-12 good). A difference of 1 point indicates significant change in function. The SPPB has been validated in patients with decompensated cirrhosis.

**3.2.3 Depression and Anxiety Symptoms:** Depression and anxiety symptoms will be obtained from the patient only. The Patient Health Questionnaire-9 (PHQ-9)<sup>53, 54</sup> and Generalized Anxiety Disorder Scale (GAD-7)<sup>55, 56</sup> will be used to measure patient mood and anxiety. The PHQ-9 is a nine-item depression scale with a total score from 0 to 27, and the GAD-7 is a seven-item anxiety scale with a total score from 0 to 21. Both of these scales are derived from the Patient Health Questionnaire, have good internal consistency and test–retest reliability as well as convergent, construct, criterion, procedural and factorial validity for the diagnosis of major depression and general anxiety disorder.

- **3.2.4 Cognitive Assessment:** Cognitive assessment will be obtained from the patient only. 3D CAM and PHES are psychometric measures of hepatic encephalopathy. They are quick, simple paper tests that are easily interpreted. They are components of the gold-standard Psychometric Hepatic Encephalopathy Score. <sup>57-60</sup>
- **3.2.5 Caregiver Burden:** Caregiver burden will be obtained from the caregiver only. The Zarit Burden Interview-12 (ZBI-12) is a validated instrument that has been utilized in various populations.<sup>61</sup> It has excellent test characteristics when compared with the long form of the ZBI, and it has been used in other studies of cirrhosis.4, <sup>62</sup>
- **3.2.6 Acute Health Care Utilization**: Health care utilization will be obtained from the patient only. In addition to patient-reported emergency room and admission data, we will use the Indiana University Health local data warehouse and the larger Indiana Network for Patient Care (INPC) to complement the utilization assessment. INPC is a large health information exchange in Indiana and provides data from all health care systems within the state. We will determine the number of emergency room visits and the number of hospitalizations within 6 months of discharge as well as associated diagnoses. As part of this, we will also be tracking admissions specific to COVID-19, due to the large impact the pandemic has had on our healthcare system. We will do that by tracking whether patients are admitted with a COVID-19 diagnosis or die of COVID-19 while enrolled in the study.
- **3.2.7 CMH Interactions:** In patients/caregivers randomized to the Cirrhosis Medical Home, we will record the numbers, timing, and types of interactions with the care coordinator (in-person, phone, video, other forms of communication). We will also record the use of interventions (e.g. care protocols, pharmacologic treatments).
- **3.2.8 Palliative Care outcomes:** Palliative care referrals will be recorded, including presence of a referral order, successful attendance at a palliative care visit, completion of advanced directives, and place of death.
- **3.3** Other Patient Measures: At baseline, we will measure age, race, gender,

level of education, income, employment, family size and household composition, height, weight, etiology of cirrhosis, liver disease severity (Child-Pugh score, 64 MELD score 65), Charlson comorbidity index, 66 medications, prior health care utilization, and reason for hospital admission.

**3.4 Other Caregiver Measures:** At baseline, we will measure age, race, gender, location (living with the patient or elsewhere), relationship to patient, and length of time caring for the patient.

The results of this study will establish the feasibility of performing a randomized trial to evaluate the efficacy of the Cirrhosis Medical Home in improving QOL for patients with decompensated cirrhosis. The next step will be to conduct a large-scale efficacy trial.

# 4.0 Eligibility Criteria

#### 4.1 Patients

#### 4.1.1 Inclusion Criteria

- Age ≥18 years
- Cirrhosis based on:
  - biopsy
  - o characteristic clinical, laboratory, and imaging findings
- Decompensated cirrhosis as denoted by any of the following:
  - o active ascites requiring paracentesis during hospitalization
  - active overt hepatic encephalopathy requiring lactulose during hospitalization
  - active hepatic hydrothorax requiring thoracentesis during hospitalization
- Poor quality of life as defined by:
   SF-36 Physical and/or Mental Component Summary scale <40 (1SD below the mean of healthy subjects)<sup>1, 40</sup>
- Discharged to home, skilled nursing facility, sub-acute rehabilitation care, or long-term acute care
- Able to be consented, either in person or through legally authorized representative
- Access to a telephone

#### 4.1.2 Exclusion Criteria

- Solid organ transplant of any organ
- History of dementing illnesses and other neurodegenerative diseases such as Alzheimer's disease, Parkinson's disease, or vascular dementia
- Unable to complete study questionnaire due to hearing loss
- Legally blind
- Pregnant or nursing
- Incarcerated

Concurrent enrollment in a related interventional research study

#### 4.2 Caregivers

# 4.2.1 Inclusion Criteria

- Age ≥18 years
- Identified caregiver of patient
- Able to be consented, either in person or through legally authorized representative
- Access to a telephone

### 4.2.2 Exclusion Criteria

- Impaired cognitive function
- Unable to complete study questionnaire due to hearing loss
- Legally blind
- Incarcerated

# 5.0 Study Design

This is a pilot, randomized controlled trial to establish the feasibility of enrollment, data collection, and outcome assessment for a future efficacy trial. Participants will be enrolled and randomized to the Cirrhosis Medical Home or usual care at the time of hospital discharge and will be followed for 6 months.

The goal of this proposal is to establish the feasibility of a randomized controlled trial comparing the Cirrhosis Medical Home to usual care in improving QOL and health care utilization of patients with decompensated cirrhosis and poor QOL. To achieve this goal, we propose a feasibility study in which we will randomize 40 patients to the Cirrhosis Medical Home or usual care, assessing QOL; physical, cognitive, and psychological symptoms; and health care utilization. Figure 1 shows the conceptual model.<sup>38</sup> We hypothesize that the Cirrhosis Medical Home will improve QOL through its effects on physical, psychological, and cognitive recovery, and that this improvement in QOL will result in decreased health care utilization.



In addition, 40 caregivers of people with cirrhosis will be enrolled in the study. They will complete the Zarit Burden Interview-12 (ZBI-12) at baseline, 3 months and 6 months. For those caregivers who care for participants who are randomized into the CMH arm, the caregivers will complete the HABC-M Caregiver assessment during their interactions with the CMH care coordinator. The HABC-M for the Caregiver is not a study outcome but is an assessment that the care coordinator uses to help guide the individualized care plan for the patient.

# 6.0 Enrollment/Randomization

Research staff will review the hepatology inpatient census each day, and eligible patients will be approached during their hospital stay. On or close to the day of hospital discharge and after obtaining informed consent, research staff will complete the Baseline Assessment and obtain baseline measurements in all enrolled subjects in both intervention and control arms. Subjects will then be randomized via a computergenerated randomization scheme into the Cirrhosis Medical Home or usual care by separate personnel who will not be involved in outcomes assessments. Research staff who are completing study assessments will be blinded to the assignment. Research staff will be trained research study personnel in the Division of Gastroenterology who will be specifically trained in the study measures. Our research assistants will be trained not to inquire about study assignments. They will be conducting structured assessments that do not provide room for qualitative interviewing that should prevent unblinding. They will not be involved in study assignments and treatment administrations. Subjects will be instructed not to discuss their therapy with the research assistants.

# 7.0 Study Procedures

**Hospital Discharge** Baseline Assessment\* Randomization **Usual** Initial Evaluation Care First Visit (≤ 72 hours) Care Plan Development Second Visit (within 2 weeks of First Visit) 6-month Interaction Period (contact at least every 2 weeks) 3 and 6 Months Outcome Measures\*

Figure 2. Study Flow

\*Assessors blinded to assignments

#### **ARM 1: Cirrhosis Medical Home**

**Initial Evaluation:** Prior to discharge, the care coordinator will review the hospital discharge plan, obtain the approval of the patient's physicians to co-manage the patient's care, and schedule a face-to-face, telephone, or virtual visit with the patient at their place of discharge. This step is important for relationship-building.

The First Visit: The care coordinator will conduct a face-to-face, telephone, or virtual visit at the patient's location (e.g. home, skilled nursing facility) within 72 hours of hospital discharge. The coordinator will assess the patient's physical, cognitive, and psychological status, and will complete a needs assessment for both the patient and family caregiver. All measures performed by the care coordinator will be used to guide the use of care protocols and development of the individualized care plan. These measures are different from the outcomes measures. The coordinator will also reconcile all medications. The Anticholinergic Cognitive Burden Scale will be completed by study staff. The coordinator will make note of scheduled and recommended appointments and will document initial and follow-up visits in the care coordination support software.

**Individualized Care Plan:** The care plan will be developed with an emphasis on coordinating services with the patient's providers. Using the assessments from the first visit, the coordinator will collaborate with the Cirrhosis Medical Home interdisciplinary team and the primary care providers to finalize the individualized care plan. This plan will be created through consultation and discussion between the care coordinator and interdisciplinary team using the assessments as guides. The assessments do not automatically trigger protocols or handouts, and there are no firm cutoffs on any of the assessments that would require any specific action. Rather, the assessments will be used to facilitate development of the care plan within the context of the patient's unique individual circumstances. The assessments will also be used to assess for response to any intervention provided, so that appropriate changes to the care plan can be made in a timely fashion. If a patient does not have a participating caregiver, then no caregiver protocols or handouts will be used. Finally, the care coordinator will schedule a second face-to-face, telephone, or virtual visit within two weeks of the first visit.

**The Second Visit:** During the second visit, the coordinator will review the individualized care plan with both the patient and the family caregiver. This process will include a) reviewing diagnoses; b) reviewing monitoring processes; c) implementation of care protocols; d) explanation of the corresponding educational handouts (patient and family caregiver); and e) connection to in-home services and community resources.

**The 6-month Interaction Period:** Follow-up includes a 6-month interaction period between the care coordinator, the patients, and the family caregivers via face-to-face visits, phone contact, email, fax, or mail. The minimum amount of contact will be every

two weeks. During these interactions, the coordinator will answer questions; collect patient and caregiver feedback; reconcile medications and discuss adherence; review appointments and care plans; have the patient and the caregiver complete the HABC Monitor to trigger the use of care protocols; and facilitate access to community resources. Additional measures, described in the schedule of events, may be repeated depending on the individualized care plan, active issues, and needs as determined by the study team. The plan will be amended through consultation and discussion between the care coordinator and interdisciplinary team using the assessments as guides. The assessments do not automatically trigger protocols or handouts and there are no firm cutoffs on any of the assessments that would require any specific action. Rather, the assessments will be used to facilitate development of the care plan within the context of the patient's unique individual circumstances. The assessments will also be used to assess for response to any intervention provided, so that appropriate changes to the care plan can be made in a timely fashion. Throughout the follow-up phase, the coordinator will work with patients, caregivers, the Cirrhosis Medical Home team, and the patient's physicians to monitor, implement, and revise the individualized care plan. Such revisions could include introducing discussions about hospice care for patients who develop indications for hospice referral during follow-up. The Cirrhosis Medical Home team and coordinator will meet weekly to discuss new patients and monitor progress. If a patient requires hospitalization, the team activates the acute care transition phase where the coordinator contacts the hospital team and provides relevant information about the patient's symptoms, as well as the patient's most updated medication list. Following any hospital discharge, the coordinator will conduct a home, telephone, or virtual visit within 72 hours to reconcile medications and coordinate the post-discharge care plan. At the end of 6 months, all patients will be transitioned to receive full care by their primary care and specialty physicians.

#### **ARM 2: Usual Care**

Prior to hospital discharge, the care coordinator will identify the primary care and/or hepatology provider of patients in the usual care group and will ensure follow up appointments at the time of hospital discharge. The coordinator will compose and send a letter to the primary care and/or hepatology provider summarizing the patient's diagnosis, hospital course, discharge medications, and the plan of follow-up care. If the patient does not already have a primary care or hepatology provider, the coordinator will work with the patient to identify a new provider. Subjects in this group will receive no further intervention.

# **Outcome Assessment (Both Arms)**

Outcome measures will be obtained by blinded research staff from all enrolled subjects at baseline, 3 months, and 6 months. Baseline assessments will be completed in the hospital at the time of enrollment. Outcomes at 3 and 6 months will be completed in person. If participants are not able to attend in person, measures that can be performed remotely will be done via phone or videoconference.

# 8.0 Study Personnel

#### 8.1 Research Staff

**8.1.1. Recruitment Staff/Assessors:** Trained research staff from the Division of Gastroenterology will be trained to administer the study measures in Section 3. They will recruit patients, obtain informed consent, complete the Baseline Assessment and measurements at the time of enrollment. They will be blinded to the study assignment as detailed in Section 6. They will also complete outcomes assessments at 3 and 6 months.

**8.1.2. Randomization Staff:** A separate member of the research team will be responsible for randomization so that the outcomes assessors will be blinded to the assignment.

### 8.2 Care Coordinator

The coordinator is a registered nurse whose scope of practice includes health coaching, case management, community organization, and nursing care. The coordinator will conduct home visits; collaborate with the interdisciplinary team; communicate with the patient's physicians; conduct root-cause analysis for unplanned acute care; implement individualized care plans; and monitor the care plans' effectiveness. The coordinator will be supervised by the interdisciplinary team. This person will conduct face to face, telephone, or virtual visit with those in the intervention arm in the hospital, within 72 hours of discharge, and again within 2 weeks (the first and second visits). They will meet with the CMH interdisciplinary team weekly throughout the study to review patients. They will assess patients using the several instruments detailed in the schedule of events, which will be used to help develop individualized care plans and which will be used to guide specific care protocols. They will interact with study participants at least every 2 weeks during the 6-month follow-up period. For those randomized to usual care, they will help ensure follow-up after discharged as detailed in Section 7, but will not have any further contact with study participants. The care coordinator will not perform any of the outcomes assessments. The coordinator will be trained in all study procedures and instruments.

# 8.3 CMH Interdisciplinary Team

The Cirrhosis Medical Home support team will consist of two hepatologists (Drs. Orman and Desai), a geriatrician with expertise in collaborative care (Dr. Boustani), a health services researcher (Dr. Fowler), and a pharmacist (Dr. Campbell). The team will meet weekly with the care coordinator. Dr. Orman will be accessible to the coordinator through phone or pager at all times. The team will supervise the care coordinator and ensure appropriate care.

# 9.0 Data Safety Monitoring

This is a minimal risk study and not a drug treatment trial. As such, adverse events are expected to be minimal in both number and nature. However, all such events or other subject problems/complications will be reported in accordance with federal, state, local, and university guidelines.

# 10.0 Study Withdrawal/Discontinuation

Participants who choose to withdraw from the study will do so by contacting the study coordinator or Dr. Orman directly at 317-278-1630. This information will be given to participants as part of the informed consent process and ongoing communication between participants and study staff.

### 11.0 Statistical Considerations

This is a pilot trial for feasibility and effect size estimation. The plan is to enroll 40 total patients and randomize in 1:1 ratio to the Cirrhosis Medical Home and usual care. As a pilot trial, the study is not powered to test efficacy, but is designed to generate preliminary data to support a larger future trial. The sample size of 40, enrolled over 9 months (see study timeline in section 13), will allow for recruitment of approximately one patient/caregiver dyad per week. Data collected from this pilot will be used to provide an estimate of intervention effect, i.e. the difference in the primary outcome measure (SF-36) between intervention and control groups. The pilot data will also provide estimates on variability in the outcome measures in this patient population. The effect and variability estimates from the pilot data will be used to power a large trial. The sample size of 40 will provide 80% probability that the 95% confidence interval for the estimated treatment difference with half-width of 0.7SD will contain the true treatment effect. The pilot sample size of 40 has also been shown to minimize the overall sample size of the pilot and the main trial together with 80% power in the main trial to detect effect sizes in the range of 0.1~0.3SD.<sup>67</sup>

# 12.0 Statistical Data Management

Primary data will be collected from conversations with the participants, both in person and via the telephone, as well as direct data capture from study instruments and the EMR and stored electronically in REDCap. The storage location will be backed up automatically, manually every day per REDCap standard procedures. Other data sources include outside medical record and lab data, data from INPC that will be stored in separate electronic files and merged with the primary data as needed. Quality assurance steps will include built in range checks and testing of database by study team prior to moving to production mode. The following quality control methods will be used:

single entry with random checks of accuracy and extraction and cleaning of data that will be used for analysis approximately every 6 months.

# **13.0 Privacy/Confidentiality Issues**

All study visits will be conducted in a private room with the door closed. Nonetheless, there is a risk of loss of confidentiality. Risks will be mitigated by conducting study visits in a private location. All paper data will be stored in locked cabinets in a locked area. Electronic data are entered and stored into a password protected database. Only authorized personnel will have access to the study data, in both paper and electronic format.

# 14.0 Follow-up and Record Retention

Subject participation will last 6 months and the entire duration of the study should take about 2 years. Study records and study data will be retained and destroyed in accordance with federal, state, local, and university guidelines.

| | Ye | ar 1 | | | Year 2 | | | |
|------------------|----|------|---|---|--------|---|---|---|
| | 1 | 2 | ვ | 4 | 1 | 2 | 3 | 4 |
| Start-up | | | | | | | | |
| Enrollment | | | | | | | | |
| Intervention | | | | | | | | |
| Outcome measures | | | | | | | | |
| Data entry | | | | | | | | |
| Data analysis | | | | | | | | |
| R01 Preparation | | | | | | | | |

### 15.0 References

- 1. Marchesini G, Bianchi G, Amodio P, et al. Factors associated with poor health-related quality of life of patients with cirrhosis. Gastroenterology 2001;120:170-8.
- 2. Healthcare Cost and Utilization Project. http://hcupnet.ahrq.gov. Accessed July 23, 2018.
- 3. D'Amico G, Garcia-Tsao G, Pagliaro L. Natural history and prognostic indicators of survival in cirrhosis: a systematic review of 118 studies. J Hepatol 2006;44:217-31.
- 4. Bajaj JS, Wade JB, Gibson DP, et al. The multi-dimensional burden of cirrhosis and hepatic encephalopathy on patients and caregivers. Am J Gastroenterol 2011;106:1646-53.
- 5. Samoylova ML, Covinsky KE, Haftek M, et al. Disability in patients with end-stage liver disease: Results from the functional assessment in liver transplantation study. Liver Transpl 2017;23:292-298.
- 6. Bajaj JS, Thacker LR, Wade JB, et al. PROMIS computerised adaptive tests are dynamic instruments to measure health-related quality of life in patients with cirrhosis. Aliment Pharmacol Ther 2011;34:1123-32.

7. Rakoski MO, McCammon RJ, Piette JD, et al. Burden of cirrhosis on older Americans and their families: analysis of the health and retirement study. Hepatology 2012;55:184-91.

- 8. Orman ES, Ghabril M, Emmett TW, et al. Hospital Readmissions in Patients with Cirrhosis: A Systematic Review. J Hosp Med 2018.
- 9. Volk ML, Tocco RS, Bazick J, et al. Hospital readmissions among patients with decompensated cirrhosis. Am J Gastroenterol 2012;107:247-52.
- 10. Agrawal K, Kumar P, Markert R, et al. Risk Factors for 30-Day Readmissions of Individuals with Decompensated Cirrhosis. South Med J 2015;108:682-7.
- 11. Stepanova M, De Avila L, Afendy M, et al. Direct and Indirect Economic Burden of Chronic Liver Disease in the United States. Clin Gastroenterol Hepatol 2017;15:759-766.e5.
- 12. Sada YH, Street RL, Jr., Singh H, et al. Primary care and communication in shared cancer care: a qualitative study. Am J Manag Care 2011;17:259-65.
- 13. Institute of Medicine Committee on the Crossing the Quality Chasm: Next Steps Toward a New Health Care S. In: Adams K, Greiner AC, Corrigan JM, eds. The 1st Annual Crossing the Quality Chasm Summit: A Focus on Communities. Washington (DC): National Academies Press (US)
  Copyright 2004 by the National Academy of Sciences. All rights reserved., 2004.
- 14. Policy and payment changes to the Medicare Physician Fee Schedule for 2015. https://www.cms.gov/Newsroom/MediaReleaseDatabase/Fact-sheets/2014-Fact-sheets-items/2014-10-31-7.html. Accessed July 24, 2018.
- 15. Callahan CM, Boustani MA, Unverzagt FW, et al. Effectiveness of collaborative care for older adults with Alzheimer disease in primary care: a randomized controlled trial. Jama 2006;295:2148-57.
- 16. Unutzer J, Katon W, Callahan CM, et al. Collaborative care management of late-life depression in the primary care setting: a randomized controlled trial. Jama 2002;288;2836-45.
- 17. Archer J, Bower P, Gilbody S, et al. Collaborative care for depression and anxiety problems. Cochrane Database Syst Rev 2012;10:Cd006525.
- 18. Vickrey BG, Mittman BS, Connor KI, et al. The effect of a disease management intervention on quality and outcomes of dementia care: a randomized, controlled trial. Ann Intern Med 2006;145:713-26.
- 19. Khan BA, Lasiter S, Boustani MA. CE: critical care recovery center: an innovative collaborative care model for ICU survivors. Am J Nurs 2015;115:24-31; quiz 34, 46.
- 20. Trauma Medical Home for Older Injured Patients: https://ClinicalTrials.gov/show/NCT03108820.
- 21. McAlister FA, Stewart S, Ferrua S, et al. Multidisciplinary strategies for the management of heart failure patients at high risk for admission: a systematic review of randomized trials. J Am Coll Cardiol 2004;44:810-9.
- 22. Feltner C, Jones CD, Cene CW, et al. Transitional care interventions to prevent readmissions for persons with heart failure: a systematic review and meta-analysis. Ann Intern Med 2014;160:774-84.
- 23. Bekelman DB, Allen LA, McBryde CF, et al. Effect of a Collaborative Care Intervention vs Usual Care on Health Status of Patients With Chronic Heart Failure: The CASA Randomized Clinical Trial. JAMA Intern Med 2018;178:511-519.
- 24. Kruis AL, Smidt N, Assendelft WJ, et al. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev 2013:Cd009437.
- 25. LaMantia MA, Alder CA, Callahan CM, et al. The Aging Brain Care Medical Home: Preliminary Data. J Am Geriatr Soc 2015;63:1209-13.

Version Date: October 4, 2021 

26. Wigg AJ, Chinnaratha MA, Wundke R, et al. A chronic disease management model for chronic liver failure. Hepatology 2015;61:725-8.

- 27. Galvin JE, Valois L, Zweig Y. Collaborative transdisciplinary team approach for dementia care. Neurodegener Dis Manag 2014;4:455-69.
- 28. Callahan CM, Boustani MA, Weiner M, et al. Implementing dementia care models in primary care settings: The Aging Brain Care Medical Home. Aging Ment Health 2011;15:5-12.
- 29. Tan ZS, Jennings L, Reuben D. Coordinated care management for dementia in a large academic health system. Health Aff (Millwood) 2014;33:619-25.
- 30. Jennings LA, Tan Z, Wenger NS, et al. Quality of Care Provided by a Comprehensive Dementia Care Comanagement Program. J Am Geriatr Soc 2016;64:1724-30.
- 31. Wigg AJ, McCormick R, Wundke R, et al. Efficacy of a chronic disease management model for patients with chronic liver failure. Clin Gastroenterol Hepatol 2013;11:850-8.e1-4.
- 32. Morando F, Maresio G, Piano S, et al. How to improve care in outpatients with cirrhosis and ascites: a new model of care coordination by consultant hepatologists. J Hepatol 2013;59:257-64.
- 33. Morales BP, Planas R, Bartoli R, et al. HEPACONTROL. A program that reduces early readmissions, mortality at 60 days, and healthcare costs in decompensated cirrhosis. Dig Liver Dis 2018;50:76-83.
- 34. Counsell SR, Callahan CM, Clark DO, et al. Geriatric care management for low-income seniors: a randomized controlled trial. Jama 2007;298:2623-33.
- 35. Bajaj JS, Riggio O, Allampati S, et al. Cognitive dysfunction is associated with poor socioeconomic status in patients with cirrhosis: an international multicenter study. Clin Gastroenterol Hepatol 2013;11:1511-6.
- 36. Berwick DM, Nolan TW, Whittington J. The triple aim: care, health, and cost. Health Aff (Millwood) 2008;27:759-69.
- 37. Frame A, LaMantia M, Reddy Bynagari BB, et al. Development and Implementation of an Electronic Decision Support to Manage the Health of a High-Risk Population: The enhanced Electronic Medical Record Aging Brain Care Software (eMR-ABC). EGEMS (Wash DC) 2013;1:1009.
- 38. Khan S, Biju A, Wang S, et al. Mobile critical care recovery program (m-CCRP) for acute respiratory failure survivors: study protocol for a randomized controlled trial. Trials 2018;19:94.
- 39. Younossi ZM, Boparai N, Price LL, et al. Health-related quality of life in chronic liver disease: the impact of type and severity of disease. Am J Gastroenterol 2001;96:2199-205.
- 40. Ware JE, New England Medical Center H, Health I. SF-36 physical and mental health summary scales: a user's manual. Boston: Health Institute, New England Medical Center, 1994.
- 41. Runyon BA. Introduction to the revised American Association for the Study of Liver Diseases Practice Guideline management of adult patients with ascites due to cirrhosis 2012. Hepatology 2013;57:1651-3.
- 42. Vilstrup H, Amodio P, Bajaj J, et al. Hepatic encephalopathy in chronic liver disease: 2014 Practice Guideline by the American Association for the Study of Liver Diseases and the European Association for the Study of the Liver. Hepatology 2014;60:715-35.
- 43. Garcia-Tsao G, Abraldes JG, Berzigotti A, et al. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology 2017;65:310-335.
- 44. Monahan PO, Alder CA, Khan BA, et al. The Healthy Aging Brain Care (HABC) Monitor: validation of the Patient Self-Report Version of the clinical tool designed to measure and

Version Date: October 4, 2021 

- monitor cognitive, functional, and psychological health. Clin Interv Aging 2014;9:2123-32.
- 45. Monahan PO, Boustani MA, Alder C, et al. Practical clinical tool to monitor dementia symptoms: the HABC-Monitor. Clin Interv Aging 2012;7:143-57.
- 46. Wang S, Allen D, Perkins A, et al. Validation of a New Clinical Tool for Post–Intensive Care Syndrome. American Journal of Critical Care 2019;28:10-18.
- 47. Harris PA, Taylor R, Thielke R, et al. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform 2009;42:377-81.
- 48. Ware JE, Jr., Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992;30:473-83.
- 49. Ware JE, Jr., Bayliss MS, Rogers WH, et al. Differences in 4-year health outcomes for elderly and poor, chronically ill patients treated in HMO and fee-for-service systems. Results from the Medical Outcomes Study. Jama 1996;276:1039-47.
- 50. Guralnik JM, Ferrucci L, Pieper CF, et al. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci 2000;55:M221-31.
- 51. Lai JC, Feng S, Terrault NA, et al. Frailty predicts waitlist mortality in liver transplant candidates. Am J Transplant 2014;14:1870-9.
- 52. Lai JC, Dodge JL, Sen S, et al. Functional decline in patients with cirrhosis awaiting liver transplantation: Results from the functional assessment in liver transplantation (FrAILT) study. Hepatology 2016;63:574-80.
- 53. Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med 2001;16:606-13.
- 54. Lowe B, Unutzer J, Callahan CM, et al. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care 2004;42:1194-201.
- 55. Kroenke K, Spitzer RL, Williams JB, et al. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med 2007;146:317-25.
- 56. Spitzer RL, Kroenke K, Williams JB, et al. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med 2006;166:1092-7.
- 57. Weissenborn K, Ruckert N, Hecker H, Manns MP. The number connection tests A and B: interindividual variability and use for the assessment of early hepatic encephalopathy. J Hepatology 1998;28(4):646-53.
- 58. Adrover R, Barrio M, Albuquerque MM, et al. Validation of the number connection test for identifying patients with minimal hepatic encephalopathy. Acta Gastroenterol Latinoam 2012;42(2):105-11.
- 59. Randolph C, Hilsabeck R, Kato A, et al. Neuropsychological assessment of hepatic encephalopathy: ISHEN practice quidelines. Liver Int 2009;29:629-35.
- 60. Weissenborn K, Ennen JC, Schomerus H, et al. Neuropsychological characterization of hepatic encephalopathy. J Hepatology 2001;34(5):768.
- 61. Higginson IJ, Gao W, Jackson D, et al. Short-form Zarit Caregiver Burden Interviews were valid in advanced conditions. J Clin Epidemiol 2010;63:535-42.
- 62. Nguyen DL, Chao D, Ma G, et al. Quality of life and factors predictive of burden among primary caregivers of chronic liver disease patients. Ann Gastroenterol 2015;28:124-129.
- 63. McDonald CJ, Overhage JM, Barnes M, et al. The Indiana network for patient care: a working local health information infrastructure. An example of a working infrastructure collaboration that links data from five health systems and hundreds of millions of entries. Health Aff (Millwood) 2005;24:1214-20.
- 64. Pugh RN, Murray-Lyon IM, Dawson JL, et al. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg 1973;60:646-9.

Version Date: October 4, 2021 

65. Kamath PS, Wiesner RH, Malinchoc M, et al. A model to predict survival in patients with end-stage liver disease. Hepatology 2001;33:464-70.

- 66. Charlson ME, Pompei P, Ales KL, et al. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis 1987;40:373-83.
- 67. Whitehead AL, Julious SA, Cooper CL, et al. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res 2016;25:1057-73.

# 16.0 Appendices

- **16.1 Schedule of Events**
- **16.2 Sample Care Plan**

Version Date: October 4, 2021 

# **16.1 Schedule of Events**

| Assessment | Baseline | Initial<br>Evaluation | First<br>Visit | Second<br>Visit | Week<br>4 | CMH Interaction* | | | | | 3<br>Month | CMH Interaction* | | | 6<br>Month | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week <sup>†</sup> | 0 | 0 | 72 hr | 2 | | 4 | 6 | 8 | 10 | 12 | | 14 | 16 | 18 | 20 | 22 | 24 | |
| Demographics | Х | | | | | | | | | | | | | | | | | |
| Height/weight | X | | | | | | | | | | | | | | | | | |
| Cirrhosis | Х | | | | | | | | | | | | | | | | | |
| etiology | | | | | | | | | | | | | | | | | | |
| MELD | X | | | | | | | | | | Χ | | | | | | | Χ |
| Child-Pugh | X | | | | | | | | | | Χ | | | | | | | Χ |
| CCI | X | | | | | | | | | | | | | | | | | |
| Medications | Χ | | Χ | X | | Х | Χ | Χ | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | |
| Reason for | X | | | | | | | | | | | | | | | | | |
| admission | | | | | | | | | | | | | | | | | | |
| SF-36 | X | | | | Χ | | | | | | X | | | | | | | Χ |
| SPPB/LFI | Х | | | | | | | | | | Х | | | | | | | Х |
| C-SSRS | | | | 1 | | / | / | / | 1 | / | | 1 | / | 1 | / | 1 | / | |
| PHQ-9 | Χ | | | | | | | | | | Х | | | | | | | Χ |
| GAD-7 | Х | | | | | | | | | | Х | | | | | | | Χ |
| PHES | X | | | | | | | | | | X | | | | | | | Χ |
| ZBI-12 | X | | | | | | | | | | X | | | | | | | Χ |
| Utilization | Х | | | | | | | | | | | | | | | | | Χ |
| HABC-M Self | | X <sup>1</sup> | | X | | Χ | Χ | Χ | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | |
| HABC-M | | X <sup>1</sup> | | Х | | Х | Х | Х | Х | Х | | Х | Х | Х | Х | Х | Х | |
| Caregiver | | | | Λ | | ^ | | ^ | ^ | ^ | | | ^ | ^ | ^ | | ^ | |
| MMSE | | X <sup>1</sup> | | 1 | | / | / | / | / | / | | 1 | / | / | 1 | / | / | |
| TUG | | X <sup>1</sup> | | 1 | | / | 1 | / | / | / | | / | / | / | / | / | / | |
| HADS | | X <sup>1</sup> | | 1 | | / | 1 | / | / | / | | / | / | / | / | / | / | |
| PEG | | X <sup>1</sup> | | 1 | | / | 1 | / | 1 | / | | 1 | / | / | 1 | 1 | / | |
| 3D CAM | | X <sup>1</sup> | | 1 | | / | / | / | / | / | | 1 | / | / | 1 | 1 | / | |
| Stroop | | X <sup>1</sup> | | 1 | | / | / | / | 1 | / | | / | / | / | / | / | / | |
| AUDIT-C | | X <sup>1</sup> | | 1 | | / | / | / | / | / | | / | / | / | / | / | / | |
| PACS | | /1 | | / | | / | / | / | / | / | | / | / | / | / | 1 | / | |

<sup>\*</sup>Interaction contacts may be in-person or via phone.

<sup>†</sup>Timing is approximate. The First Visit is within 72 hours of hospital discharge. The Second Visit is within 2 weeks of the First Visit. CMH Interactions occur a minimum of every 2 weeks.

X = required (HABC-M Caregiver only if caregiver enrolled)

/ = optional, depending on clinical circumstance

 $X^1$  = can be performed at initial evaluation or first visit

Performed by Blinded Research Staff for all enrolled subjects

Performed by CMH Care Coordinator only for those randomized to the Cirrhosis Medical Home

Patient assessments

Caregiver assessments

Abbreviations: MELD, Model for End-Stage Liver Disease; CCI, Charlson Comorbidity Index; SF-36, Short Form Survey; SPPB, Short Physical Performance Battery; LFI, Liver Frailty Index; PHQ-9, Patient Health Questionnaire; GAD-7, Generalized Anxiety Disorder;; ZBI-12, Zarit Burden Interview; HABC-M, Healthy Aging Brain Care Monitor; MMSE, Mini-Mental Status Examination; TUG, Timed Up-and-Go; HADS, Hospital Anxiety and Depression Scale; PEG, Pain, Enjoyment, General Activity Scale; 3D CAM-, Confusion Assessment Method for the ICU

Version Date: October 4, 2021 


16.2 Sample Care Plan

| Study ID #: | Age: | | | | | | | | | | Gender: |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Occupation: | Educ: | 3 m | | | 6 m | | 9 m | | | 12m | Ethnicity: |
| Instrument | 7/11 | 10/5 | 10/19 | 11/2 | 2/27 | 3/28 | 5/23 | 6/27 | 7/24 | 9/13 | Targets |
| <u>MMSE</u> | - | | | | - | | | | | - | - |
| Orientation Time | 5/5 | | | | 5/5 | | | | | 5/5 | |
| Orientation Place | 5/5 | | | | 5/5 | | | | | 5/5 | |
| Registration | 3/3 | | | | 3/3 | | | | | 3/3 | |
| Attention & | 5/5 | | | | 5/5 | | | | | 5/5 | |
| Calculation | 3/3 | | | | 3/3 | | | | | 3/3 | |
| Recall | 2/2 | | | | 2/2 | | | | | 2/2 | |
| Naming | 1/1 | | | | 1/1 | | | | | 1/1 | |
| Repetition | 3/3 | | | | 3/3 | | | | | 3/3 | |
| Comprehension | 1/1 | | | | 1/1 | | | | | 1/1 | |
| Reading | 1/1 | | | | 1/1 | | | | | 1/1 | |
| Writing | 1/1 | | | | 1/1 | | | | | 1/1 | |
| Drawing | 30 | | | | 30 | | | | | 30 | >27 |
| Total | | | | | | | | | | | |
| <u>HADS</u> | - | - | | | - | | _ | | | - | _ |
| Anxiety | 13 | 9 | | | 7 | | 0 | | | 0 | <7 |
| Depression | 7 | 2 | | | 0 | | 0 | | | 0 | <7 |
| TUG | UTC | UTC | | | UTC | | UTC | | | UTC | <9 sec |
| PEG | 4.33 | 3.33 | 2.3 | 2 | 1.66 | 2.33 | 2.66 | 2.33 | 0 | 2.33 | <4 |
| 3D CAM | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <20 |
| Stroop | | | | | | | | | | | <190 |
| HABC-SRM | - | - | - | _ | - | - | - | _ | - | - | - |
| Cognitive | 2 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <4 |
| Functional | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | <3 |
| Behavioral & Mood | 8 | 8 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | <5 |
| Total | 13 | 8 | 5 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | <14 |
| Score 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | |
| Score 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | |
| Score 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | |
| Total ACB | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | <2 |

Care Coordinator suggests implementing highlighted protocols below **Protocols**:

- 1. Cognition
- 2. Exercise
- 3. Depression
- 4. Anxiety

- 5. Physical Health
- 6. Behavioral Care
- 7. Legal and Financial
- 8. Communication
- 9. Mobility
- 10. Personal Care
- 11. Sleep Disturbance
- 12. Pain
- 13. Stress
- 14. Acute Care Reduction/DELIRIUM
- 15. Medication Adherence
- 16. Ascites/Edema
- 17. Hepatic Encephalopathy
- 18. Alcohol and Substance Use Disorder Protocol

#### Care Plan:

- 1. Counseling (Prognosis & Natural History)
- 2. Enhancing Knowledge
- 3. Brain Exercises / Cognitive Rehabilitation
- 4. Physical Exercise / Physical Rehabilitation
- 5. Time-Off Caregiving Tasks (minimum of 8 hours per week)
- 6. Belonging to Support Group
- 7. Counseling (Coping with Disease Disability)
- 8. Respite Care
- 9. Medication Adherence Support
- 10. Referral or starting Cognitive Behavioral Therapy
- 11. Referral or starting Problem Solving Therapy
- 12. Referral for Family Therapy
- 13. Referral for Home Health Care Services
- 14. Referral to Adult Day Care
- 15. Referral for Driving Evaluation / Rehab
- 16. Recommend Residing in Assisted Living
- 17. Referral to Elder Low Attorney
- 18. Referral to Elder Abuse Agency Investigation
- 19. Referral for Guardianship
- 20. Counseling for Advance Directives
- 21. Prescribe ChEI
- 22. Prescribe Antidepressants
- 23. Prescribe Vascular Burden Reduction
- 24. Reduce Anticholinergic Burden
- 25. Prescribe Anxiolytics
- 26. Prescribe Sleep Medication
- 27. Prescribe Other